CLINICAL TRIAL: NCT05103800
Title: Investigation of the Effect of White Noise Listening on Pain and Comfort During Invasive
Brief Title: Investigation of the Effect of White Noise Listening on Pain and Comfort During Invasive Interventions in Newborns
Acronym: IEWNLPCDIIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Tugba Todi̇l, Lecturer, Batman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BatmanU
Record Dates: First submitted 2021-09-06; First posted 2021-11-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Pain, Acute; Child Behavior; Newborn
Keywords: Child Health and Nursing; Pain; Newborn; Comfort
MeSH Terms: conditions — Acute Pain; Child Behavior; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Babies in the control group will not listen to any sound during the invasive procedures, the procedure will be recorded with a camera, and at the end of the study, the camera images will be watched by two experts in the field and the pain and comfort scale will be filled.
- Experimental group (Experimental): During the invasive interventions, the white noise prepared by the researcher for the babies in the experimental group will be started to be listened to 5 minutes before the start of the intervention and will be listened to for 5 more minutes during and after the intervention. At the same time, the procedure will be recorded with a camera. At the end of the study, the camera images will be watched by two experts in the field. comfort scale will be filled.
  Interventions: Behavioral: invasive interventions

INTERVENTIONS:
Behavioral: invasive interventions — listening the white noise during the invasive interventions
  Other Names: white noise
  Arms: Experimental group

SUMMARY:
Comfort, distress and the absence of pain can be described as free from anxiety, somewhat enjoyable and ease (peaceful) situation. The child health and disease nurse should come up with physiological problems of the baby, increase the comfort degree to reduce the stress level of the baby and ensure improvement in the baby's location. This research was experimentally designed to investigate the effect of the baby's own intrauterine heart sound on pain and comfort during the invasive procedures applied to the healthy born babies in the delivery units of the Batman Gynecology and Pediatrics Hospital.

The research will be performed by selecting samples in a simple random sampling method from the babies who born healthy and timely in the normal vaginal way. The number of samples will be determined by power analysis method after pilot study. The previously white noise will have listened to the babies in experimental group and will be recorded by camera during invasive interventions and the pain and comfort scale will be applied. The scales will be applied to the control group let them without listening White noise but also will be recorded with camera and thus the data will be collected. A nurse working in the unit will perform invasive interventions, later two specialists will watch video records and so the pain and comfort scales will be filled.

No study on this subject was found in the international literature review. Based on the need to fill this gap in the literature, it seems that the study will contribute to the field of child health and diseases nursing.

DETAILED DESCRIPTION:
Comfort can be defined as the absence of distress and pain, free from anxiety, somewhat pleasurable and relaxed (peaceful) situation. Providing comfort and calmness of the child, relieving pain and distress are applications in the physical field of comfort theory. Nursing interventions applied in newborns are an integral component of professional nursing care to increase patient comfort level. The child health and diseases nurse should provide solutions to the baby's physiological problems, increase the comfort level to reduce the baby's stress level, and improve the baby's environment.

Many invasive attempts are applied to the newborn baby after birth without being discharged from the hospital. These applications, which cause tissue destruction, are painful for babies. This study was designed as experimentally in order to examine the effect of listening white noise on pain and comfort during the invasive procedure applied to healthy babies in the delivery room of Batman Training and Research Hospital. The hypotheses for this research were determined as follows:

H10: Listening to white noise in newborn babies during an invasive intervention does not affect the baby's pain.

H11: Listening to white noise in newborn babies during an invasive intervention reduces the baby's pain.

H20: Listening to white noise in newborn babies during an invasive intervention does not affect the comfort of the baby.

H21: Listening to white noise in newborn babies during an invasive intervention increases the comfort of newborn babies.

In the literature review, studies were found in which attempts were made to alleviate the interventional pain of the newborn using one or more of the sensory stimuli such as visual, auditory, tactile, taste and smell. In the treatment of pain in the newborn; various alternative and complementary treatments are used such as positioning, swaddling, rocking, holding, kangaroo care applied by mother/father, massage, acupressure, reiki application, pacifier, sweet solutions (sucrose, glucose), breastfeeding, listening to the mother's voice, singing, lullaby, aromatherapy and, smelling familiar scents. In the literature review, the application of white noise listening to the baby during an invasive procedure or otherwise is limited.

In this thesis, it is aimed to increase the quality of care provided, to listen to white noise during the invasive interventions applied to the baby, to observe the effect on the baby's pain and comfort, to reduce the pain and to increase the comfort of the baby, and to be a source for similar studies.

RESOURCE SUMMARY The International Organization for Pain Studies (ISAP) has defined the most valid concept of pain today, which is a universal experience and has been tried to be explained by human beings for centuries. According to this organization, pain, is always subjective as it is an unpleasant nature that accompanies or can be defined by existing or potential tissue damage. Although the most reliable indicator in pain assessment is the patient's own expression, different pain diagnosis methods are used when evaluating pediatric patients who have difficulty in expressing their pain. Providing comfort and calmness of the child, relieving pain and distress are applications in the physical field of comfort theory. Providing this aspect of comfort is possible with pain assessment and interventions for it.

Comfort, which is a word of French origin and is defined as the comfort that makes daily life easier in the dictionary meaning, in nursing; it consists of the process of diagnosing the comfort needs of the patient, family or society, taking precautions for their needs, evaluating the basic comfort level and the comfort level after the application. According to Kolcaba, comfort is "an expected result with a complex structure in physical, psycho-spiritual, social and environmental integrity related to helping the individual's needs, providing peace and overcoming problems". Kolcaba, as a result of her analytical studies on the use of the concept of comfort in the nursing discipline; stated that it is a positive, holistic, multidimensional, theoretically definable and practical concept. The concept of comfort according to the holistic view; it is the satisfaction of basic human needs in order to find relief, find peace and overcome problems.

After nurses started to give care systematically, they started to use various concepts; concepts such as comfort (relaxation), care, and communication formed the basis of theory development studies. Comfort, which is a concept traditionally associated with the art of nursing, is an individual and holistic concept. It has been reported in the literature that the nurses provide strength, care, support, encouragement and assistance through comfort and comfort measures.

The concept of comfort has been used frequently in neonatal intensive care units and newborn babies in recent years. In studies, it is stated that one of the most important factors affecting the recovery rate is comfort. Kolcaba et al. emphasized that comfort has the effect of increasing the benefit and cost ratios, and the level of patient satisfaction. Increasing the patient comfort level by applying nursing interventions in newborns is an integral component of professional nursing care. The child health and diseases nurse should provide solutions to the baby's physiological problems, increase the comfort level to reduce the baby's stress level, and improve the baby's environment.

In the literature review, studies were found in which attempts were made to alleviate the interventional pain of the newborn using one or more of the sensory stimuli such as visual, auditory, tactile, taste and smell. In the treatment of pain in the newborn various alternative and complementary treatments are used, such as; positioning, swaddling, rocking, holding, kangaroo care made by mother/father, massage, acupressure, reiki application, pacifier, sweet solutions (sucrose, glucose), breastfeeding, listening to the mother's voice, singing, lullaby, aromatherapy and smelling familiar smells.

Aslan recommends the use of non-pharmacological methods to minimize the pain that occurs during heel blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Babies who were born by normal vaginal delivery
* Babies who were born in the delivery room of Batman Training and Research Hospital

Exclusion Criteria:

* Congenital anomalies
* Cranial hemorrhage
* Who need oxygen support
* Who have sepsis or suspected sepsis

Ages: 5 Minutes to 3 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Newborn Comfort Behavior Scale (COMFORTneo Behavior Scale) | 6 months
  Newborn Comfort Behavior Scale is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. It was stated that the lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6, and the highest score is 30. High scores indicate that the baby is not comfortable and needs interventions to provide comfort. In addition, a score of 4-6 on the numerical evaluation scales indicates moderate pain and a score of 7-10 indicates severe pain and distress.

SECONDARY OUTCOMES:
Neonatal Infant Paint Scale | 6 months
  The Neonatal Infant Paint Scale is measured by evaluating five behavioral groupings (facial expression, crying, movements of arms and legs, alertness) and a physiological indicator (breathing pattern). Total pain scores range from 0-7. (0-2 = mild to no pain, 3-4 = mild to moderate pain, >4 = severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba TODIL, Principal Investigator — Cukurova University
Locations (1):
- Çukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No